CLINICAL TRIAL: NCT03504059
Title: School-based Behavioural Intervention to Face Obesity and Promote Cardiovascular Health Among Spanish Adolescents: a Cluster-randomized Controlled Trial
Brief Title: School-based Behavioural Intervention to Face Obesity and Promote Cardiovascular Health Among Spanish Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: SHE Foundation (Other); Centro Nacional de Investigaciones Cardiovasculares Carlos III (Unknown); Fundació La Marató de TV3 (Other); Obra social La Caixa (Unknown)
Responsible Party: Principal Investigator, Rosa M Lamuela-Raventós, Associate Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 369/C/2016
Record Dates: First submitted 2018-01-09; First posted 2018-04-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Cardiovascular Health; Diabetes Mellitus
Keywords: Obesity; Cardiovascular Health; Diabetes; Adolescents; Physical Activity; Diet; School-Based
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): The usual educational program is applied
- Short Intervention (Active Comparator): A two-year specially designed educational program is applied. This program aims to encourage a healthy lifestyle through gamification, including diet education, physical activity and self esteem.
  Interventions: Behavioral: Short-term educational program
- Long Intervention (Active Comparator): A four-year specially designed educational program is applied. This program aims to encourage a healthy lifestyle through gamification, including diet education, physical activity and self esteem.
  Interventions: Behavioral: Long-term educational program

INTERVENTIONS:
Behavioral: Long-term educational program — Comprehensive educational school-based intervention in adolescents on cardiovascular health, including obesity/adiposity and metabolic profiles, through classroom intervention, and complementary intervention in the family setting, at school and on teachers.
  Arms: Long Intervention
Behavioral: Short-term educational program — Comprehensive educational school-based intervention in adolescents on cardiovascular health, including obesity/adiposity and metabolic profiles, through classroom intervention, and complementary intervention in the family setting, at school and on teachers.
  Arms: Short Intervention

SUMMARY:
Background and objective:

There is an alarming increase in obesity and unhealthy lifestyles in adolescents. This issue threatens to have a highly negative health and socioeconomic impact in the near future. The only way to tackle this epidemic is to implement effective preventive strategies able to positively impact on youth lifestyle behaviours. The school is the most appropriate environment for such an intervention. The main objective of this study is to evaluate the efficacy of a comprehensive educational school-based intervention in adolescents on cardiovascular health, including obesity/adiposity and metabolic profiles. The project consortium constitutes a unique framework of research groups at the forefront of novel and successful approaches aiming to healthier behaviours and dietary habits.

Methodology:

A cluster-randomized controlled trial involving 24 secondary schools in Spain will be carried out. Schools will be 1:1:1 randomized to receive a short-term (2-year) or a long-term (4-year) comprehensive educational program, or to receive the usual curriculum (control). Participants will be evaluated at baseline, and after 2 and 4 years with the following: weight scale, circumference measuring tape, bioelectrical impedance, dual energy X-ray absorptiometry, sphygmomanometer, blood analysis, saliva and urine analysis, accelerometers, and questionnaires. The primary outcome is the change in obesity and other health parameters from baseline to year 2 and 4, as assessed by the Ideal Cardiovascular Health score. Secondary outcomes include the change in adiposity, anthropometry and body composition parameters, physical activity and dietary habits, polyphenol and carotenoid intake, metabolomics and attitudes. Participants will be measured again when they reach 20 years old.

Expected results:

The investigators expects to show that a school-based educational intervention induces favorable lifestyle changes and improves cardiovascular health among Spanish adolescents, including obesity/adiposity and metabolic profiles. If successful, this strategy could be widely adopted having a meaningful effect on obesity and cardiovascular health promotion. Additionally, associations between health parameters and bioactive dietary compounds intake and metabolic profiles will be stablished.

ELIGIBILITY:
Inclusion Criteria:

* • Any student studying the first academic year of secondary school (Enseñanza Secundaria Obligatoria, ESO) in the selected high schools.

Exclusion Criteria:

* No exclusion criteria.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1326 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the composite ICH score of adolescents from baseline to year 2 and 4 | 2 and 4 years
  The ICH score measures cardiovascular health and includes 7 components:
  - Behaviors factors:
  1. No smoking
  2. Being physically active
  3. Good nutritional habits
  4. Normal weight
     - Health factors:
  5. Normal blood pressure
  6. Normal cholesterol level
  7. Normal glucose levels To meet the complete definition of ideal cardiovascular health, an individual would need to meet the ideal levels of all 7 components.

SECONDARY OUTCOMES:
Changes in body mass index from baseline to year 2 and 4 | 2 and 4 years
  Change in body mass index (kg/m^2), calculated after measure weight (kg) and height (meter).
Changes in waist circumference from baseline to year 2 and 4 | 2 and 4 years
  Change in waist circumference (cm) measured in triplicate
Changes in percentage of body fat from baseline to year 2 and 4 | 2 and 4 years
  Change in total adiposity measured by bioelectrical impedance (percentage of fat).
Changes in distribution of body fat from baseline to year 2 and 4 | 2 and 4 years
  Change in adiposity distribution measured by dual energy X-ray absorptiometry, that calculate total body fat, regional fat, including android, gynoid, visceral and lean mass.
Changes in dietary habits from baseline to year 2 and 4 | 2 and 4 years
  To evaluate the association between food and nutrient intake and changes in adiposity parameters. To assess changes in diet and adherence to the Mediterranean diet a validated Food Frequency Questionnaire (FFQ) (Tresserra-Rimbau et al., 2013) will be used. A shorter FFQ (Children's Eating Habits Questionnaire - Food Frequency Questionnaire (CEHQ-FFQ) (Lanfer et al., 2011; Bel-Serrat et al. 2014)) will also be used to analyze dietary patterns.
Changes in attitudes about eating from baseline to year 2 and 4 [ Time Frame: 2 and 4 years | 2 and 4 years
  To evaluate the relationship between changes in attitudes and changes in adiposity parameters. A validated questionnaire will be used to assess attitudes about eating (Lima-Serrano et al., 2012).
Changes in polyphenol consumption from baseline to year 2 and 4 | 2 and 4 years
  Dietary polyphenol (PP) intake will be estimated from FFQ and data from the PP content in foods, obtained from the Phenol-explorer data base. With this methodology, it can obtain an estimation of total PP intake by each individual and different PP classes. For the determination of phenolics and their metabolites in human urine, will be used solid-phase extraction and ultra-HPLC coupled to mass spectrometry (Martinez-Huelamo et al., 2015).
Changes in carotenoids consumption from baseline to year 2 and 4 | 2 and 4 years
  Carotenoids and retinol consumption will be also estimated from the longer FFQ. Total energy and micronutrient intake will be obtained using the Food Processor Nutrition and Fitness Software (ESHA Research, Salem, OR).
Changes in energy and nutrients consumption from baseline to year 2 and 4 | 2 and 4 years
  Total energy and micronutrient intake will be obtained from a validated Food Frequency Questionnaire (Tresserra-Rimbau et al., 2013) using the Food Processor Nutrition and Fitness Software.
Changes in metabolomics from baseline to year 2 and 4 | 2 and 4 years
  To evaluate the effect of the intervention on metabolism through a metabolomic approach. Urine and salivary samples will be collected to perform a metabolomics analysis in order to evaluate metabolic changes due to educational intervention on dietary and physical activity habits. Liquid chromatography coupled to quadrupole time of-flight mass spectrometry (HPLC-q-TOF) will be used for such analysis which is able to measure thousands of metabolites simultaneously from only minimal amounts of sample. Data mining analysis will be performed using XCMS-R package. The preprocessed data obtained by XCMS in negative and positive ionization will be separately exported to SIMCA 13.0.3 software (Umetrics) to perform unsupervised and supervised multivariate analysis to detect metabolic changes among groups.
Changes in physical activity from baseline to year 2 and 4 | 2 and 4 years
  To study the association between changes in physical activity and changes in adiposity parameters . Actigraph wGT3X-BT accelerometers that allow the registration of the amount and intensity of physical activity will be used during 7 days per evaluation time-point. To complete this information a diary with questions about the type of physical activity performed during the 7 days will be collected. A validated questionnaire will be also used to assess physical activity habits (Barbosa et al., 2007).
Changes in sedentary habits from baseline to year 2 and 4 | 2 and 4 years
  To study the association between changes in sedentary habits and changes in adiposity parameters. Information on sedentary time from Actigraph wGT3X-BT accelerometers will be taken into account. In addition, we will measure sedentary leisure time spent with the computer/console/TV /mobile (ENSE 2012).
Changes in attitudes towards abuse substances from baseline to year 2 and 4 | 2 and 4 years
  The attitudes towards abuse substances will be assessed by a validated questionnaire (Lima-Serrano et al., 2013). An additional questionnaire will be used to assess self-efficacy (Markham et al., 2009).
Changes in smoking habits from baseline to year 2 and 4 | 2 and 4 years
  Validated questionnaires will be used to assess smoking status itself, and in its immediate environment (Moreno et al., 2012 Lana, 2010).
Changes in perception of the self-image from baseline to year 2 and 4 | 2 and 4 years
  A questionnaire to assess the perception of the self-image will be used to obtain a pattern of individual acceptance with his/her figure (Stunkard et al., 1990).
Changes in self-esteem from baseline to year 2 and 4 | 2 and 4 years
  Self-esteem will be assessed using validated questionnaire (Rajmil et al., 2003).
Changes in emotional eating from baseline to year 2 and 4 | 2 and 4 years
  Emotional eating will be assessed using validated questionnaire (Jauregui-Lobera et al., 2014)
Changes in mood from baseline to year 2 and 4 | 2 and 4 years
  Self-efficacy will be assessed using a validated questionnaire (Vázquez Fernández et al., 2013).
Evaluation of the shorter vs. longer educational intervention effectiveness by comparison of 2 and 4 year results on all outcomes | 4 years
  The effectiveness of a shorter vs. longer educational intervention program (2 and 4 year) will be assessed by comparison of final (4 year) results on all proposed outcomes.
Cardiovascular score validation | 4 years
  The BEWAT score, which includes the assessment of Blood pressure, Exercise, Weight, Alimentation (fruit and vegetables) and Tobacco consumption, will be also derived. This simple and non-invasive score (score from 0 to 15 points) will be validated against the ICH score, and will serve for future studies in adolescents.
Changes in the composite ICH score of adolescents from baseline to adulthood | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Lamuela-Raventós, PhD, Principal Investigator — University of Barcelona; Gloria Santos-Beneit, PhD, Principal Investigator — SHE Foundation; Juan M Fernández Alvira, PhD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III; Valentín Fuster, PhD, MD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III
Locations (3):
- Spain (3):
  - School of Pharmacy. University of Barcelona., Barcelona, Barcelona
  - Fundación SHE, Barcelona, Barcelona
  - Centro Nacional de Investigaciones Cardiovasculares Carlos III, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martinez-Gomez J, Bodega P, Santos-Beneit G, de Cos-Gandoy A, Beneito-Dura M, de Miguel M, Tresserra-Rimbau A, Ruiz-Leon AM, Estruch R, Lamuela-Raventos RM, Moreno LA, Fernandez-Alvira JM, Fernandez-Jimenez R. Trajectories of adherence to an obesogenic dietary pattern and changes in diet quality, food intake, and adiposity during adolescence. Nutr J. 2025 Mar 7;24(1):35. doi: 10.1186/s12937-025-01102-y. PMID 40055723
- [Derived] Arancibia-Riveros C, Dominguez-Lopez I, Laveriano-Santos EP, Parilli-Moser I, Tresserra-Rimbau A, Ruiz-Leon AM, Sacanella E, Casas R, Estruch R, Bodega P, de Miguel M, de Cos-Gandoy A, Martinez-Gomez J, Santos-Beneit G, Fernandez-Alvira JM, Fernandez-Jimenez R, Lamuela-Raventos RM. Unlocking the power of polyphenols: A promising biomarker of improved metabolic health and anti-inflammatory diet in adolescents. Clin Nutr. 2024 Aug;43(8):1865-1871. doi: 10.1016/j.clnu.2024.06.023. Epub 2024 Jun 25. PMID 38964203
- [Derived] Bodega P, Santos-Beneit G, de Cos-Gandoy A, Moreno LA, de Miguel M, Orrit X, Tresserra-Rimbau A, Martinez-Gomez J, Ramirez-Garza SL, Laveriano-Santos EP, Arancibia-Riveros C, Estruch R, Lamuela-Raventos RM, Fernandez-Jimenez R, Fernandez-Alvira JM. Clustering of lifestyle behaviors and adiposity in early adolescents in Spain: findings from the SI! Program for Secondary Schools. BMC Public Health. 2023 Aug 12;23(1):1535. doi: 10.1186/s12889-023-16461-6. PMID 37568128
- [Derived] Santos-Beneit G, Fernandez-Alvira JM, Tresserra-Rimbau A, Bodega P, de Cos-Gandoy A, de Miguel M, Ramirez-Garza SL, Laveriano-Santos EP, Arancibia-Riveros C, Carral V, Orrit X, Rodriguez C, Carvajal I, Haro D, Peyra C, Martinez-Gomez J, Alvarez-Benavides A, Estruch R, Lamuela-Raventos RM, Fernandez-Jimenez R, Fuster V. School-Based Cardiovascular Health Promotion in Adolescents: A Cluster Randomized Clinical Trial. JAMA Cardiol. 2023 Sep 1;8(9):816-824. doi: 10.1001/jamacardio.2023.2231. PMID 37531100
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Fernandez-Jimenez R, Santos-Beneit G, Tresserra-Rimbau A, Bodega P, de Miguel M, de Cos-Gandoy A, Rodriguez C, Carral V, Orrit X, Haro D, Carvajal I, Ibanez B, Storniolo C, Domenech M, Estruch R, Fernandez-Alvira JM, Lamuela-Raventos RM, Fuster V. Rationale and design of the school-based SI! Program to face obesity and promote health among Spanish adolescents: A cluster-randomized controlled trial. Am Heart J. 2019 Sep;215:27-40. doi: 10.1016/j.ahj.2019.03.014. Epub 2019 Apr 10. PMID 31277052